CLINICAL TRIAL: NCT01140932
Title: Electroretinographic Changes in Healthy Young Men Before and After Induction of Glucose Intolerance by Glucocorticoids Treatment, Hyperphagia and Lack of Exercise
Brief Title: The Electroretinogram in Healthy and Glucose Intolerant Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Michael Larsen, MD, DMsc, Glostrup University Hospital,Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Kappelgaard, ERG
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Electroretinography
Keywords: Retina; Electroretinography; Diabetes Mellitus; Glucose Intolerance; Physiology
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — Prednisolone; Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Medical and behavioural intervention
  Interventions: Drug: Prednisolone; Behavioral: Lifestyle change

INTERVENTIONS:
Drug: Prednisolone — 12 days of corticosteroids treatment (prednisolone 37,5 mg/day)
  Other Names: Prednisolon DAK, Nycomed, Zurich, Switzerland
Behavioral: Lifestyle change — High calorie diet (130 % of recommended daily energy intake) and relative physical inactivity (no exercise and at least 8 hours of rest/day)
  Other Names: Behavioral regimen

SUMMARY:
The purpose is to investigate the electroretinogram (ERG) in young, healthy men in the normoglycaemic and hyperglycaemic state before and after intervention with corticosteroids treatment, high calorie diet and exercise restraint.

DETAILED DESCRIPTION:
The subjects will be fasting from midnight the day before the experiment. Standard procedures (including pupil dilation, dark adaptation, and local anaesthetics) are carried out to allow the ERG to be obtained. After electrophysiology, the subject will be clamped at a plasma glucose level of 10 mM (~180 mg/dL) and after a stabilisation period the ERG protocol is repeated.

Each subject is examined twice on two different days. The first day the subjects are normoglycaemic in the morning (first examination) and hyperglycaemic (clamped to 10 mM) throughout the second examination. The second day subjects are also normoglycaemic and hyperglycaemic but shows up after 7-12 days of daily intake of prednisolone, high calorie diet, and exercise restraint.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians without type 2 diabetes mellitus
* Normal OGTT (75 g glucose dissolved in 250 mL water) according to WHO's criteria
* BMI 20-30
* Haemoglobin > 8,0 mM

Exclusion Criteria:

* Nephropathy (s-creatinin > 130 µM or albuminuria)
* Relatives (parents or sibling with T2DM)
* Medical treatment which cannot be paused for 12 hours

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
ERG | 12 days
  Characteristics of the scotopic ERG at normo-/hyperglycaemia before vs. after prednisolone treatment

SECONDARY OUTCOMES:
Retinal Vessel Caliber | 12 days
  Measurement of retinal vessel caliber from fundus photographs before and after treatment with glucocorticoids.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Larsen, MD, DMsc, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Copenhagen University Hospital at Glostrup, Copenhagen, Copenhagen, Denmark